CLINICAL TRIAL: NCT02500121
Title: A Randomized, Double-blinded, Phase II Study of Maintenance Pembrolizumab Versus Placebo After First-Line Chemotherapy in Patients With Metastatic Urothelial Cancer: Hoosier Cancer Research Network GU14-182
Brief Title: Testing the PD-1 Inhibitor Pembrolizumab as Maintenance Therapy After Initial Chemotherapy in Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCRN GU14-182
Record Dates: First submitted 2015-07-08; First posted 2015-07-16 (Estimated); Results first posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: Pembrolizumab; PD-1 Inhibitor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm A (Placebo Comparator): Commercially available normal saline will be used as the placebo. No active placebo drug will be mixed with the normal saline. Treatment will continue, in the absence of prohibitive toxicities or disease progression, for up to 24 months.
  Interventions: Other: Placebo
- Experimental Arm B (Experimental): Pembrolizumab, 200mg IV every 3 weeks. Treatment will continue, in the absence of prohibitive toxicities or disease progression, for up to 24 months.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Other: Placebo — Normal saline
  Arms: Control Arm A
Drug: Pembrolizumab — Pembrolizumab, 200mg IV every 3 weeks until progressive disease, unacceptable toxicity, or for up to 24 months
  Arms: Experimental Arm B

SUMMARY:
This is a multi-institutional, randomized, placebo controlled, double-blinded phase II trial of maintenance pembrolizumab versus placebo after first-line chemotherapy in patients with metastatic urothelial cancer who have achieved at least stable disease on first-line chemotherapy.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

Eligible subjects will be 1:1 randomized to placebo (Control Arm A) and pembrolizumab (Experimental Arm B). Stratification factors for randomization: presence of visceral metastatic disease (lung, liver, or bone or other organs vs. lymph node only) at the time of initiation of first-line chemotherapy, and response to first-line chemotherapy (CR/PR vs. SD. Subjects who progress on placebo will be assessed to determine if they are eligible to cross over to unblinded treatment with pembrolizumab.

INVESTIGATIONAL TREATMENT:

For Control Arm A, commercially available normal saline will be used as the placebo. No active placebo drug will be mixed with the normal saline.

For Experimental Arm B, pembrolizumab (or placebo), 200 mg intravenous infusion (IV) every 3 weeks for up to 12 months, or until progressive disease (PD) or unacceptable toxicity.

The following required laboratory values must be obtained within fourteen days prior to registration for protocol therapy:

Hematopoietic:

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥8.5 g/dL

Renal:

* Creatinine ≤1.5x ULN OR
* Measured or calculated creatinine clearance ≥30 mL/min for subject with creatinine levels >1.5x institutional ULN
* GFR can also be used in place of creatinine or CrCl

Hepatic:

* Serum total bilirubin ≤ 1.5 X ULN OR
* Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subject with liver metastases

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN. If subject is on anticoagulant therapy, PT or PTT must be within therapeutic range of intended use of anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status (PS) of ≤ 1 within fourteen days of registration for protocol therapy.
* Histological or cytological evidence of urothelial cancer of the bladder, urethra, ureter, or renal pelvis. Differentiation with variant histologies (e.g., squamous cell differentiated) will be permitted provided that the predominant histology is urothelial carcinoma.
* Metastatic and/or unresectable (cT4b) disease
* Must have achieved an objective response (CR/PR) or stable disease (SD) after 4 to 6 cycles of standard first-line platinum-based chemotherapy for mUC (e.g., as per NCCN guidelines). Able to commence study treatment within 2 to 6 weeks of receiving last dose of first-line chemotherapy.
* All subjects must have adequate archival tissue available prior to registration (i.e., at least 20 unstained slides or paraffin block). If acceptable archival tissue is not available, the subject must be willing to consent to providing a core or excisional biopsy for research prior to registration for protocol therapy. If archival tissue is not available and there are no sites amenable to biopsy, enrollment must be discussed with the sponsor-investigator on a case by case basis.
* Female subjects of childbearing potential must have a negative serum pregnancy within three days prior to registration for protocol therapy
* Sexually active, pre-menopausal women of childbearing potential must be willing to use an adequate method of contraception or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study drug. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > one year.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* More than one line of prior chemotherapy for metastatic or locally advanced disease, with the following exception:

  * Prior neoadjuvant/adjuvant chemotherapy will not count as line of therapy if completed greater than 12 months prior to initiation of chemotherapy regimen for metastatic or unresectable disease.
* Current or past participation in a study of an investigational agent or using an investigational device within four weeks of registration for protocol therapy.
* A diagnosis of immunodeficiency or is receiving treatment with systemic steroid therapy or any other form of immunosuppressive therapy within seven days prior to registration for protocol therapy.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within two weeks prior to registration for protocol therapy. Note: If the subjects have undergone major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting protocol therapy.
* A known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* A known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to registration for protocol therapy and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least seven days prior to registration for protocol therapy.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has evidence of active, non-infectious pneumonitis.
* Has a history of interstitial lung disease.
* An active infection requiring systemic therapy.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening period through 120 days after the last dose of protocol therapy.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). Examples include nivolumab, MPDL3280, etc.
* A known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* A known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Receipt of a live vaccine within 30 days prior to registration for protocol therapy.
* Unresolved toxicity (i.e., > Grade 1 or above baseline) due to previously administered agents. Exception includes: subjects with ≤ Grade 2 neuropathy are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, M.D., Study Chair — Hoosier Cancer Research Network
Locations (28):
- United States (28):
  - University of Arizona at Dignity Health St. Joseph's, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - IU Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Community Healthcare System, Munster, Indiana
  - University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University: Siteman Cancer Center, St Louis, Missouri
  - GU Cancer Research Network, LLC, Omaha, Nebraska
  - The John Theuer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galsky MD, Mortazavi A, Milowsky MI, George S, Gupta S, Fleming MT, Dang LH, Geynisman DM, Walling R, Alter RS, Kassar M, Wang J, Gupta S, Davis N, Picus J, Philips G, Quinn DI, Haines GK 3rd, Hahn NM, Zhao Q, Yu M, Pal SK. Randomized Double-Blind Phase II Study of Maintenance Pembrolizumab Versus Placebo After First-Line Chemotherapy in Patients With Metastatic Urothelial Cancer. J Clin Oncol. 2020 Jun 1;38(16):1797-1806. doi: 10.1200/JCO.19.03091. Epub 2020 Apr 9. PMID 32271672
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm A | Experimental Arm B
Started | 53 | 55
Crossover to Pembrolizumab | 27 (Only subjects that progressed on the control arm were eligible to participate in the crossover portion of the trial.) | 0 (Not applicable for the experimental arm.)
Completed (All subjects that) | 26 | 29
Not Completed | 27 | 26
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 26 | 24

BASELINE CHARACTERISTICS:
Population: One patient randomly assigned to placebo was excluded from the analysis because of inconsistent receipt of pembrolizumab rather than placebo during the initial several cycles of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm A | Experimental Arm B | Total
Number analyzed (Participants) | 52 | 55 | 107
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 87] | 68 [41 to 83] | 66 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 42 | 39 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 46 | 50 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 52 | 55 | 107
Presence of Visceral Metastatic Disease at time of Initiation of First Line Chemotherapy [Count of Participants; unit: Participants] — Subjects on this study were stratified by presence of visceral metastatic disease at the time of initiation of fire-line chemotherapy. Visceral metastatic disease is defined by disease in the lung, liver, or bone.
  Participants | 32 | 39 | 71
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead.
  Measured at baseline.
  Participants
    ECOG 0 | 23 | 22 | 45
    ECOG 1 | 29 | 33 | 62
Cycles of First-Line Chemotherapy [Median (Inter-Quartile Range); unit: cycles] | 6 [4 to 6] | 6 [4 to 6] | 6 [4 to 6]
Best Response to First Line Chemotherapy [Count of Participants; unit: Participants] — Subjects were stratified by their response to first line chemotherapy (Complete or Partial Response vs Stable Disease).
  Participants
    Complete Response/Partial Response | 36 | 40 | 76
    Stable Disease | 16 | 15 | 31
Cisplatin based First Line Chemotherapy [Count of Participants; unit: Participants] — Whether first-line therapy regimen was cisplatin based.
  Participants | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Measured at the time from randomization to death or progression, depending on which occurs first, as per immune-related RECIST (irRECIST). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Calculated after a median follow-up time of 12.9 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 52 | 55
months | 3.0 [2.7 to 5.5] | 5.4 [3.1 to 7.3]

2. Secondary Outcome: 6-month PFS as Per irRECIST
Description: Probability that subjects remain alive and progression free at 6 months post randomization per irRECIST criteria. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Six months after randomization
Population: as for baseline characteristics
Measure: Number; unit: probability
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 52 | 55
probability | 0.2551 | 0.4101

3. Secondary Outcome: Number of Subjects With Adverse Events as a Measure of the Safety and Tolerability of Pembrolizumab
Description: Percentage of subjects with treatment-emergent grade 3-4 toxicities, as per Common Terminology Criteria for Adverse Events (CTCAE) v 4.0
Time Frame: Every 3 weeks beginning with C1D1 for up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 52 | 55
percentage of participants | 38 | 59

4. Secondary Outcome: Objective Response Rate (ORR) Assessment of Subjects on Maintenance Pembrolizumab vs Placebo
Description: The objective response rate is the percentage of all subjects with confirmed PR or CR according to RECIST, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment)
  Complete Response per RECIST 1.1 is defined as the disappearance of all target and non-target lesions and the reduction in size of any pathologic lymph nodes to <10mm in the absence of the appearance of any new lesions.
  Partial Response per RECIST 1.1 is defined by at least a 30% decrease in the sum of the diameters of target lesions when compared to baseline, no equivocal progression of non-target disease and no appearance of new lesions.
Time Frame: Response assessed every 12 weeks from the date of randomization to the date of documented disease progression or date of death, whichever occurs first, assessed for up to a maximum of 104 weeks (24 months)
Population: Only subjects with measureable disease per RECIST 1.1 at baseline were considered assessable for this endpoint. 10 subjects on Arm A and 12 subjects on Arm B were enrolled on the study with a complete response to previous therapy at baseline. One patient randomly assigned to placebo was excluded from the analysis because of inconsistent receipt of pembrolizumab rather than placebo during the initial several cycles of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 42 | 43
percentage of participants | 10 | 23

5. Secondary Outcome: ORR Assessment of Subjects Receiving Pembrolizumab After Progressing on Placebo
Description: as for outcome 4
Time Frame: Every 12 weeks from the first treatment on the crossover to the date of documented disease progression, per irRECIST 1.1, assessed for up to a maximum of 104 weeks (24 months)
Measure: Number; unit: percentage of participants
Groups:
- Crossover: Arm A subjects that experienced progressive disease per RECIST 1.1 and opted to participate in the crossover portion of the trial. Subjects received pembrolizumab (200mg) every 3 weeks for up to 24 months.
Arm/Group | Crossover
Number analyzed (Participants) | 27
percentage of participants | 22

6. Secondary Outcome: Median Overall Survival (OS) Time in Subjects Treated With Pembrolizumab vs Placebo
Description: Median time from randomization until death from any cause in subjects treated with pembrolizumab vs placebo.
Time Frame: From randomization until death from any cause. Reported after a median follow-up of 12.9 months.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 52 | 55
months | 18.7 [11.4 to NA] — upper limit has not been achieved due to insufficient number of participants with events. | 22 [12.9 to NA] — upper limit has not been achieved due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) up to 25 months.
Groups:
- Arm A: Commercially available normal saline will be used as the placebo. No active placebo drug will be mixed with the normal saline. Treatment will continue, in the absence of prohibitive toxicities or disease progression, for up to 24 months. Placebo: Normal saline
- Arm B: Pembrolizumab, 200mg IV every 3 weeks. Treatment will continue, in the absence of prohibitive toxicities or disease progression, for up to 24 months.
  Pembrolizumab: Pembrolizumab, 200mg IV every 3 weeks until progressive disease, unacceptable toxicity, or for up to 24 months
Arm/Group | Arm A | Arm B | Crossover
All-Cause Mortality (participants affected / at risk) | 12/53 | 24/55 | 14/27
Serious Adverse Events (participants affected / at risk) | 10/53 | 25/55 | 6/27
Other Adverse Events (participants affected / at risk) | 50/53 | 51/55 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=53) | Arm B (N=55) | Crossover (N=27)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HEMATOMA (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
STROKE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
AUTOIMMUNE DISORDER (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
EDEMA LIMBS (General disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
FEVER (General disorders) | 0 (0) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (3) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULAR DISORDERS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=53) | Arm B (N=55) | Crossover (N=27)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (10) | 4 (6) | 4 (4)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 1 (1) | 2 (2)
AGITATION (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 10 (17) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 8 (12) | 12 (18) | 3 (3)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
ANAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 19 (34) | 17 (42) | 7 (17)
ANOREXIA (Metabolism and nutrition disorders) | 7 (7) | 9 (10) | 5 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2) | 2 (2)
ASCITES (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5) | 12 (21) | 2 (3)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (8) | 9 (10) | 2 (3)
BLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (5) | 3 (3) | 1 (2)
BLURRED VISION (Eye disorders) | 2 (2) | 6 (6) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
CHILLS (General disorders) | 2 (2) | 5 (9) | 2 (2)
CHOLESTEROL HIGH (Investigations) | 1 (1) | 0 (0) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (4) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CONFUSION (Psychiatric disorders) | 1 (1) | 3 (4) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 11 (12) | 13 (19) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 15 (15) | 7 (18)
CREATININE INCREASED (Investigations) | 13 (23) | 16 (40) | 5 (10)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (5) | 3 (5) | 2 (3)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 10 (11) | 20 (32) | 5 (7)
DIZZINESS (Nervous system disorders) | 9 (10) | 7 (8) | 2 (2)
DRY EYE (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 3 (3) | 1 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 14 (16) | 5 (7)
EDEMA FACE (General disorders) | 1 (1) | 0 (0) | 1 (1)
EDEMA LIMBS (General disorders) | 5 (6) | 9 (10) | 3 (4)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
EYE DISORDERS (Eye disorders) | 1 (3) | 2 (2) | 1 (2)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 3 (5) | 0 (0)
FATIGUE (General disorders) | 20 (29) | 21 (34) | 7 (11)
FEVER (General disorders) | 6 (7) | 5 (7) | 3 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (13) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
FLOATERS (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (3)
GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (2) | 0 (0) | 4 (5)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 1 (1)
HEADACHE (Nervous system disorders) | 5 (5) | 6 (10) | 3 (3)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HEMATOMA (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 9 (14) | 9 (18) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 (20) | 11 (64) | 7 (12)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 5 (6) | 5 (9) | 2 (2)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 11 (15) | 9 (20) | 5 (8)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 6 (6) | 6 (12) | 5 (11)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (6) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 6 (8) | 9 (20) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (2) | 3 (3) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 5 (6) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 3 (5) | 11 (12) | 1 (2)
IRRITABILITY (General disorders) | 1 (1) | 0 (0) | 0 (0)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LOCALIZED EDEMA (General disorders) | 1 (1) | 2 (2) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 8 (18) | 17 (35) | 2 (3)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7) | 1 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (5)
NAUSEA (Gastrointestinal disorders) | 10 (10) | 9 (15) | 4 (9)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 2 (8) | 0 (0)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 6 (9) | 6 (7) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (14) | 3 (3)
PARESTHESIA (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
PARONYCHIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 3 (4) | 4 (6) | 1 (2)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6 (8) | 9 (9) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 7 (8) | 7 (11) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
PROLAPSE OF INTESTINAL STOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (7) | 13 (19) | 2 (3)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (24) | 2 (2)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 3 (3) | 3 (4) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (13) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 5 (7) | 2 (3) | 2 (5)
URINARY FREQUENCY (Renal and urinary disorders) | 3 (3) | 3 (6) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 10 (13) | 2 (3)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
VOMITING (Gastrointestinal disorders) | 2 (3) | 9 (18) | 2 (5)
WEIGHT GAIN (Investigations) | 1 (1) | 1 (1) | 0 (0)
WEIGHT LOSS (Investigations) | 2 (3) | 2 (2) | 3 (3)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (3) | 5 (13) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 4 (4) | 2 (2)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC DISORDERS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN - CARDIAC (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
ENDOCRINE DISORDERS (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 3 (3) | 2 (2)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1) | 0 (0)
GALLBLADDER PAIN (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GENITAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
GGT INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
HEMOGLOBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HOT FLASHES (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 5 (5) | 1 (1)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 0 (0)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1)
IMMUNE SYSTEM DISORDERS (Immune system disorders) | 0 (0) | 1 (1) | 1 (4)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INR INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
LIP INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (6) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
MOVEMENTS INVOLUNTARY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NECK EDEMA (General disorders) | 0 (0) | 1 (2) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 3 (3) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PENILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PENILE PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PHOTOSENSITIVITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
SERUM AMYLASE INCREASED (Investigations) | 0 (0) | 1 (2) | 0 (0)
SKIN HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 5 (5) | 0 (0)
URINARY URGENCY (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
VASCULAR DISORDERS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
WATERING EYES (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02500121/Prot_SAP_000.pdf